CLINICAL TRIAL: NCT03014102
Title: Recombinant Human Thrombopoietin for Mobilization of Peripheral Blood Progenitor Cells for Autologous Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hongnan Mo (Other)
Responsible Party: Sponsor-Investigator, Hongnan Mo, Attending Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LC2016B03
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Thrombocytopoietin; Hematopoietic Stem Cell Mobilization; Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Thrombopoietin

ARMS (2):
- TPOqd (Experimental): Recombinant Human Thrombopoietin 300U/kg/d ih quaque die, day-3/-2/-1 before mobilization
  Interventions: Drug: Recombinant Human Thrombopoietin
- TPOqod (Active Comparator): Recombinant Human Thrombopoietin 300U/kg/d ih qua altera die, day-3/-1/+2 before mobilization
  Interventions: Drug: Recombinant Human Thrombopoietin

INTERVENTIONS:
Drug: Recombinant Human Thrombopoietin — Recombinant human Thrombopoietin is a full length glycosylated molecule identical to endogenous Thrombopoietin.

SUMMARY:
The purpose of this study is to determine whether recombinant human thrombopoietin are effective in peripheral blood progenitor cells mobilization for autologous transplantation.

ELIGIBILITY:
Inclusion Criteria:

* a histologically confirmed diagnosis of Hodgkin's disease, non-Hodgkin's lymphoma, or selected high-risk solid tumors that are planned to receive autologous peripheral blood progenitor cell transplantation
* Eastern Cooperative Oncology Group performance status of 0 - 2.

Exclusion Criteria:

* abnormal liver function (aminotransferase or bilirubin levels 2 times upper limit of normal), leukopenia (white blood cell count 3000/L), or a history of platelet or other disorders associated with a bleeding diathesis
* a history of thromboembolic disease, coronary heart disease,stroke, arrhythmias, central nervous system metastases,or other organ system diseases or abnormalities that might predispose individuals to treatment-related complications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
the average number of cluster of differentiation 34 positive cells/kg | up to 24 months
  To evaluate the effect of combining various treatment schedules of recombinant human thrombopoietin with granulocyte colony stimulating factor on the mobilization of peripheral blood progenitor cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Mo H, Liu P, Qin Y, He X, Han X, Yao J, Su W, Zhang S, Tang L, Zhao F, Gui L, Yang S, Yang J, Zhou S, Zhang Z, Shi Y. Recombinant human thrombopoietin prior to mobilization chemotherapy facilitates platelet recovery in autologous transplantation in patients with lymphoma: Results of a prospective randomized study. Chronic Dis Transl Med. 2021 Jun 24;7(3):190-198. doi: 10.1016/j.cdtm.2021.05.003. eCollection 2021 Sep. PMID 34505019